CLINICAL TRIAL: NCT00171431
Title: The Effect of Tegaserod on Patterns of Flow in the Small Bowel of Patients With Irritable Bowel Syndrome (IBS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early in May 2006 due to low patient enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919AUS33
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Constipation Predominant; Irritable Bowel Syndrome (IBS-C)
Keywords: IBS-C; female
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Evaluation of the effect of tegaserod treatment on small intestinal motility and flow pattern in female IBS-C patients.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 and older
* IBS-C patients diagnosed on the basis of Rome II criteria
* Ability to comply with the requirements of the entire study

Exclusion Criteria:

* Evidence of structural abnormality of the gastrointestinal tract or disease/conditions.
* Patients with previous gastrointestinal surgery other than appendectomy or cholecystectomy.
* Evidence of cathartic colon or a history of laxative use, that in the investigator's opinion is consistent with severe laxative dependence such that the patient is likely to require or use laxatives during the study

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of tegaserod on motility and small intestinal flow patterns after meal in female patients with IBS-C
by using Multiple Intraluminal Impedance

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States